CLINICAL TRIAL: NCT02254876
Title: Effectiveness of NeuroMuscular Taping in a Population of Post Stroke Hemiplegic Patients Suffering From Painful Shoulder Syndrome - Randomized Controlled Trial (RCT)
Brief Title: Effectiveness of NeuroMuscular Taping on Painful Hemiplegic Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, paolo pillastrini, Associate Professor and President of Baccaluareate Course in Physiotherapy, University of Bologna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4496/2013
Record Dates: First submitted 2014-09-29; First posted 2014-10-02 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Hemiplegia
Keywords: Stroke; Hemiplegia; Painful shoulder Syndrome; NeuroMuscolar Taping
MeSH Terms: conditions — Hemiplegia; Stroke

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard physical therapy program (Active Comparator): Standard physical therapy program is delivered for four rehabilitation sessions for a period of about 45 minutes each.
  Interventions: Other: Standard physical therapy program
- NeuroMuscular Taping (NMT) (Experimental): NeuroMuscular Taping is delivered in addiction to the "Standard Treatment" for four rehabilitation sessions. The sessions were spaced apart about five days to ensure the optimum adhesion of the NMT.
  Interventions: Other: Standard physical therapy program; Other: NeuroMuscular Taping (NMT)

INTERVENTIONS:
Other: Standard physical therapy program — Standard physical therapy program in this study involves joint health and passive mobility at the level of the shoulder girdle and upper limb affected by Painful Shoulder Syndrome associated with the modulation of hypertonic muscle groups.
Other: NeuroMuscular Taping (NMT) — The NeuroMuscular Taping (NMT) consists of the application on the skin of an adhesive tape with a particular structure to elastic waves and with characteristics comparable to those cutaneous. Because of these characterises it allows activation of endogenous analgesic, structural and muscular support, vascular and lymphatic activation.
  In this study the NMT is applied with decompressive mode on Pectoralis Major, Deltoids, Supraspinatus.
  Arms: NeuroMuscular Taping (NMT)

SUMMARY:
Painful Shoulder Syndrome is a frequent complication after stroke occurring in between 5% and 84% of patients, often having a strong impact on their well-being and resulting in delays achieving rehabilitative objectives.

The aim of the study is to demonstrate the effectiveness of Neuromuscular Taping in a population of post-stroke hemiplegic patients suffering from painful shoulder syndrome with respect to pain, spasticity and range of motion.

DETAILED DESCRIPTION:
The study will use two groups according to the methodology of Randomized Controlled Trials. Both components of the two groups were treated by four rehabilitation sessions defined as "standard". This involves joint health and passive mobility for the glenohumeral and scapulothoracic joints for a period of about 45 minutes each.

The patients of the sample group underwent the application of the NeuroMuscular Taping (NMT) before each rehabilitative session. The control group was addressed exclusively to the "standard" treatment. The sessions were spaced apart about five days to ensure the optimum adhesion of NMT.

The results were evaluated by administering rating scales for pain (VAS) and spasticity (Modified Ashworth Scale). The ROM was evaluated using the manual goniometer. The outcomes (Pain, Spasticity, ROM) were assessed at base line, before and after each treatment session and at 1 month follow up.

ELIGIBILITY:
Inclusion Criteria:

* Right or left hemiplegia resulting from an ischemic or hemorrhagic stroke
* Painful Shoulder Syndrome, with pain at rest and during functional movement of the shoulder girdle
* Spasticity with an Ashworth score greater than or equal to 1.

Exclusion Criteria:

* Flaccidity
* Thermoalgesic sensitivity deficits
* Previous surgery to the shoulder
* Cognitive impairment
* Taking anti-inflammatory drugs and/or muscle relaxants during the course of the trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-09; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Pain | Before and after each treatment session and at 1 month follow up
  The investigators assessed this outcome with a Visual Analogue Scale (VAS).

SECONDARY OUTCOMES:
Spasticity | Before and after each treatment session and at 1 month follow up
  The investigators assessed this outcome with the Modified Ashworth Scale.
ROM | Before and after each treatment session and at one month follow up.
  The investigators assessed this outcome using manual goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Pillastrini, Principal Investigator — University of Bologna
Locations (1):
- Policlinico S.Orsola-Malpighi, Bologna, Emilia-Romagna, Italy

REFERENCES:
- [Background] Camerota F, Galli M, Cimolin V, Celletti C, Ancillao A, Blow D, Albertini G. Neuromuscular taping for the upper limb in Cerebral Palsy: A case study in a patient with hemiplegia. Dev Neurorehabil. 2014 Dec;17(6):384-7. doi: 10.3109/17518423.2013.830152. Epub 2013 Oct 2. PMID 24087981
- [Background] Murie-Fernandez M, Carmona Iragui M, Gnanakumar V, Meyer M, Foley N, Teasell R. [Painful hemiplegic shoulder in stroke patients: causes and management]. Neurologia. 2012 May;27(4):234-44. doi: 10.1016/j.nrl.2011.02.010. Epub 2011 Apr 22. Spanish. PMID 21514698
- [Background] Smith M. Management of hemiplegic shoulder pain following stroke. Nurs Stand. 2012 Jul 4-10;26(44):35-44. doi: 10.7748/ns2012.07.26.44.35.c9191. PMID 22876427